CLINICAL TRIAL: NCT05049772
Title: Investigation of the Effects of Telerehabilitation-based Motor Imagery Training in Patients With Nonspecific Low Back Pain: A Randomized Controlled Study.
Brief Title: Telerehabilitation-based Motor Imagery in Nonspecific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Collaborators: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Muhammed Zahid Uz, Lecturer, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6385-GOAEK
Record Dates: First submitted 2021-09-08; First posted 2021-09-20 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2024-07

CONDITIONS: Motor Imagery
Keywords: non-specific low back pain; telerehabilitation; motor imagery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Telerehabilitation-based motor imagery group (Experimental): Behavioral: Telerehabilitation-based motor imagery group Participants in the Telerehabilitation-based motor imagery group will imagine for the lumbar region exercises (e.g. bridges, knee-to-chest stretches, pelvic tilts) in the sessions in home using the study audio-video motor imagery script for 2 times per week; 30 min per day for 10 weeks. Phone calls will be performed for support and as a reminder for the assessment (after one week). In addition, the participants will be given stabilization exercises In addition, the participants will be given stabilization exercises for 10 weeks for 40 minutes, 2 days a week.
  Interventions: Behavioral: Telerehabilitation-based motor imagery training; Behavioral: Stabilization exercises group
- Stabilization Exercises group (Active Comparator): Behavioral: Stabilization Exercises group An exercise program consisting of lumbar stabilization exercises for the participants will be planned for the pelvic ring muscles to develop the neutral lumbar spine. Co-contraction of the transversus abdominus muscle and the multifidus muscle will form the basis of the exercises. Stabilization exercises will be given for 10 weeks for 40 minutes, 2 days a week.
  Interventions: Behavioral: Stabilization exercises group
- Healthy control group (No Intervention): no specific intervention

INTERVENTIONS:
Behavioral: Telerehabilitation-based motor imagery training — 10 weeks of motor imagery training and stabilization exercises.
  Arms: Telerehabilitation-based motor imagery group
Behavioral: Stabilization exercises group — 10 weeks of stabilization exercises.
  Arms: Stabilization Exercises group; Telerehabilitation-based motor imagery group

SUMMARY:
Low back pain is a common problem in society and causes loss of workforce. Its lifetime prevalence reaches 80% and annual hospital admission rates in the adult population reach 15%.Most studies on motor imagery suggested the effects of motor imagery are related to neuroplastic changes in the brain. Studies have shown that similar brain regions are activated during motor imagery and real movement. However, the level of evidence about the effect of motor imagery on autonomic functions is limited. Today, interest in telerehabilitation has increased due to the Covid-19 pandemic.

The aim of this study is to examine the effects of telerehabilitation-based motor imagery training in patients with non-specific low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Those who can read and write
* Patients who have not undergone surgery
* Those with a body mass index less than 30 m2/kg
* To have sufficient computer knowledge to participate in the study or to have a relative who can help in this regard
* Having a computer and active internet connection at home

Exclusion Criteria:

* Medically uncontrolled and uncooperative patients
* Patients who have undergone surgery to the lumbar region
* History of falling in the last 6 months
* Those with serious orthopedic, vascular, neurological, psychiatric problems affecting balance
* Active malignancy
* Pregnancy
* Having severe vision and hearing problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-10-08 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-16 (Actual)

PRIMARY OUTCOMES:
Feasibility of the methods - minimum recruitment rate | through Study Completion, an Average of 10 Months
  A minimum recruitment rate of 10 participants per month will be accepted as feasiable.
Feasibility of the methods - minimum retention rate | through Study Completion, an Average of 10 Months
  A target retention rate of 80% will be accepted as feasiable
Feasibility of the methods - minimum adherence rate | through Study Completion, an Average of 10 Months
  A target minimum adherence rate of 70% of the overall practice sessions will be accepted as feasiable.
Feasibility of the methods - adverse events | through Study Completion, an Average of 10 Months
  A record sheet was prepared for possible adverse events during the tests and intervention. It includes information about seriousness, expectedness, severity, causality, time, duration of the event and clinical action taken. The numbers of adverse events will be reported

SECONDARY OUTCOMES:
Kinesthetic and Visual Imagery Questionnaire | Change from Baseline at 10 Weeks
  The Kinesthetic and Visual Imagery Questionnaire-Short Form consists of 10 movements in total, measuring 5 visual and 5 kinesthetic visualization skills, developed to determine the extent to which individuals visualize and feel the imagined movements. The questionnaire is not a self-report scale, but is administered with an evaluator. All movements are evaluated in the sitting position. Higher scores indicate greater visual clarity or intensity of sensations.
Movement Imagery Questionnaire-Revised | Change from Baseline at 10 Weeks
  The Movement Imagery Questionnaire-Revised assesses visual and kinesthetic movement imagery ability and is comprised of four visual and four kinesthetic items. Each item entails performing a movement, visually or kinesthetically imaging that movement and then rating the ease or difficulty of generating that image on a 7-point scale from 1 = very hard to see/feel to 7 = very easy to see/feel. Higher scores indicate higher visual or kinesthetic movement imagery ability.
Oswestry Disability Questionnaire, | Change from Baseline at 10 Weeks
  The Oswestry Disability Questionnaire, which allows the patient to self-evaluate, is used to evaluate the limitations that patients compare in daily life. The total score ranges from 0 to 100, and a high score indicates an increased level of disability.
International Physical Activity Questionnaire | Change from Baseline at 10 Weeks
  It is grouped as Low (Category 1), Medium (Category 2), Very active (Category 3). Calculation is made on a weekly basis as MET level x minutes of activity.
VISUAL ANALOGUE SCALE | Change from Baseline at 10 Weeks
  Visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.
Wechsler Adult Intelligence Scale- Revised | Change from Baseline at 10 Weeks
  In this test, the patient is asked to repeat the digits read to him, one second apart, in the same order backwards, starting from the last. The test starts with a two-digit number sequence, and when repeated correctly, one digit is increased and continues until the seventh sequence of eight numbers. The patient must repeat at least one of the two sequences of numbers of the same length in the correct order in order to progress in the test. Scoring is based on the total number of correct and repetitions.
d2 Attention-Tests | Change from Baseline at 10 Weeks
  The test form consists of 14 lines, each with 47 marked letters. There are 16 letters "p" and "d" marked with one, two, three or four lowercase lines in each line. The patient is asked to find and cross out the letters "d" with only two signs. For each line, the patient is given 20 seconds.
Trail Making Test | Change from Baseline at 10 Weeks
  The Trail Making test consists of two parts. In Part A, the patient is asked to put together the circles with numbers in the correct order, which are scattered on the test form. In Part B, the patient is asked to combine the circles, which are scattered on the test form and contain both numbers and letters, in the correct order (1-A, 2-B, 3-C).
Pittsburg Sleep Quality Index | Change from Baseline at 10 Weeks
  The Pittsburg Sleep Quality Index evaluates sleep quality over the past month. 19 of the 24 questions included in the Pittsburg Sleep Quality Index are self-report questions. Five questions are answered by the spouse or a roommate. The 18 items participating in the scoring are grouped into 7 component scores. Each item is evaluated over 0-3 points. The sum of the 7 component scores gives the overall Pittsburg Sleep Quality Index score.
SF-36 Short Fotm | Change from Baseline at 10 Weeks
  The SF-36 has a total of 8 sub-components: physical function, physical role limitation, pain, general perception of health, vitality (energy), social function, emotional role limitation, and mental health. The answers to the questions answered by the participants are scored between 0-100. A high score indicates a good quality of life, and a low score indicates a poor quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Bilge Kara, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided